CLINICAL TRIAL: NCT06357793
Title: Evaluation of Work Productivity and Activities of the Relative Living With a Patient With Fibromyalgia Syndrome
Brief Title: Evaluation of Work Productivity and Activities of the Fibromyalgia Patients' Relatives
Status: Not yet recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: camsakuraftr
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Fibromyalgia; Work Productivity; Quality of Life; Pain, Chronic
Keywords: fibromyalgia; work productivity and activity impairment; quality of life
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fibromyalgia: The revised 2016 American College of Rheumatology (ACR) FM diagnostic criteria going to be use to diagnose FM participants group. Their relatives will fill out the WPAI:GH Questionnaire and World Health Organization Quality of Life (WHOQOL).
- control: Healthy participants' relatives will fill out the WPAI:GH Questionnaire and World Health Organization Quality of Life (WHOQOL).

SUMMARY:
Patients suffering from fibromyalgia (FM) are challenged by symptoms such as chronic pain, fatigue, sleep disturbance and emotional distress. Patients diagnosed with fibromyalgia can also negatively affect the relatives they live with due to their existing complaints. It is possible that their relatives accompanying them may lose their workforce due to untreated pain complaints and frequent hospital admissions. The main purpose of our study is to examine whether there is any impact on the working life of the people they live with and whether there is a decrease in their work productivity.

DETAILED DESCRIPTION:
This cross-sectional study will evaluate FM patients and their relatives, who are in paid full- or part time employment at the time of the assessment. The study protocol doesn't require any medical intervention. Fibromyalgia severity will be assessed with the fibromyalgia impact questionnaire (FIQ). Evaluation of patient relatives' work productivity and activities will be made with the Work Productivity and Activity Impairment questionnaire: General Health (WPAI:GH). Analyzes will be completed with a group of healthy controls in the study.

ELIGIBILITY:
Inclusion Criteria:

Study Group:

Must live together with a patient diagnosed with FM 18-65 years old Must work in a full-time/part-time job

Control Group:

Must live with a healthy relative 18-65 years old Must work in a full-time/part-time job

Exclusion Criteria:

Must live alone Not having a full-time/part-time job

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The revised 2016 American College of Rheumatology (ACR) FM diagnostic criteria were used to diagnose FM. Our study group participants have to live with FM patients. Also they have to work in a full or part-time job.
Sampling Method: Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Work Productivity and Activity of Fibromyalgia Patients' Relatives | 1 day
  Work Productivity and Activity Impairment questionnaire

SECONDARY OUTCOMES:
Quality of life Fibromyalgia Patients' Relatives | 1 day
  World Health Organization Quality of Life questionnaire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salaffi F, Di Carlo M, Farah S, Mariani C, Fulginei S, Martino GP, Sarzi-Puttini P. A cross-sectional research on female workers examining the loss of productivity caused by mild, moderate and severe fibromyalgia. Clin Exp Rheumatol. 2022 Jun;40(6):1151-1158. doi: 10.55563/clinexprheumatol/hut4ft. Epub 2022 Jun 8. PMID 35699070
- [Background] Neumann L, Buskila D. Quality of life and physical functioning of relatives of fibromyalgia patients. Semin Arthritis Rheum. 1997 Jun;26(6):834-9. doi: 10.1016/s0049-0172(97)80027-3. PMID 9213382
- [Background] Tutoglu A, Boyaci A, Koca I, Celen E, Korkmaz N. Quality of life, depression, and sexual dysfunction in spouses of female patients with fibromyalgia. Rheumatol Int. 2014 Aug;34(8):1079-84. doi: 10.1007/s00296-014-2944-z. Epub 2014 Jan 9. PMID 24402006